CLINICAL TRIAL: NCT03619252
Title: Pneumococcal Vaccination of Multiple Myeloma Patients on Novel Agents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Minsk Scientific-Practical Center for Surgery, Transplantation and Hematology (Other Government)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Principal Investigator, Ihar Iskrou, Head of Cell Transplant Division, Minsk Scientific-Practical Center for Surgery, Transplantation and Hematology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HEM-3_2
Record Dates: First submitted 2018-07-17; First posted 2018-08-07 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Multiple Myeloma; Pneumococcal Infection; Febrile Neutropenia; Pneumococcal Pneumonia
MeSH Terms: conditions — Multiple Myeloma; Pneumococcal Infections; Febrile Neutropenia; Pneumonia, Pneumococcal | interventions — Vaccination; Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vaccination group (Experimental): Patients receiving novel agents (Bortezomib/Lenalidomide/Ixazomib/Daratumumab) and enrolled in vaccination by pneumococcal conjugate vaccine (PCV13): 3 doses with 1 month interval, and fourth dose planned to be administered 6 months later.
  Interventions: Biological: Vaccination with pneumococcal conjugate vaccine (PCV13)
- Standard prophylaxis (Active Comparator): Patients receiving novel agents (Bortezomib/Lenalidomide/Ixazomib/Daratumumab) and receiving standard institutional antibacterial prophylaxis by Levofloxacin 500 mg daily during the median four cycles of treatment by novel agents
  Interventions: Drug: Standard Antibacterial Prophylaxis

INTERVENTIONS:
Biological: Vaccination with pneumococcal conjugate vaccine (PCV13) — Vaccination with pneumococcal conjugate vaccine - PCV13 (Prevnar 13/Prevenar 13, Pfizer Inc) containing saccharides from serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F individually conjugated to nontoxic diphtheria cross-reactive material. Vaccination regimen: 3 doses monthly, with a booster dose 6 months later.
  Arms: Vaccination group
Drug: Standard Antibacterial Prophylaxis — Levofloxacin 500 mg once daily during the median four cycles of treatment by novel agents.
  Arms: Standard prophylaxis

SUMMARY:
Multiple myeloma is an incurable blood cancer of plasma cells that occurs in older individuals. Novel agents (proteasome inhibitors, immunomodulatory agents) have substantially improved the overall response rates, progression-free survival and overall survival in patients with multiple myeloma. Patients with multiple myeloma are at high risk of developing life-threatening Streptococcus pneumoniae infections, while clinical efficacy and safety of conjugate pneumococcal vaccines in multiple myeloma patients receiving novel agents have not been studied before. The main aim of this study is to assess the clinical efficacy and safety of 13-valent pneumococcal conjugate vaccine in multiple myeloma patients treated with novel agents.

DETAILED DESCRIPTION:
Multiple myeloma is an incurable blood cancer of plasma cells that occurs in older individuals with a median age at diagnosis of 69 years and a median overall survival of 6-7 years [Kumar S.K., et al. Leukemia, 2014; Rollig C., et al. Lancet., 2015]. Over the past years novel agents have been introduced into clinical practice, showing improved overall response rates, progression-free survival and overall survival in patients with multiple myeloma. The main classes of novel agents include proteasome inhibitors, immunomodulatory agents and monoclonal antibodies. These agents are typically used in doublet or triplet regimens that include a chemotherapeutic drug and/or corticosteroid.

Streptococcus pneumoniae (pneumococcus) is a cause of worldwide morbidity and mortality. Patients with multiple myeloma are at high risk of developing life-threatening Streptococcus pneumoniae infections due to chemotherapy-associated immunosuppression. Vaccination is an important preventive strategy against infections caused by S. pneumoniae. In the past, the 23-valent pneumococcal polysaccharide vaccine was recommended. However, polysaccharide vaccines have limited efficacy in cancer and hematology patients, because of the decreased T- and B-cell responses. Clinical efficacy and safety of conjugate pneumococcal vaccines in multiple myeloma patients receiving novel agents have not been studied before.

In this study the investigators wish to study the effect of vaccination with 13-valent pneumococcal conjugate vaccine in multiple myeloma patients treated with novel agents (proteasome inhibitors and immunomodulatory drugs). The main aim of this study is to assess the clinical efficacy and safety of 13-valent pneumococcal conjugate vaccine in multiple myeloma patients treated with novel agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven diagnosis of multiple myeloma
* Patients must be enrolled in treatment with novel agents (Bortezomib/Lenalidomide/Ixazomib/Daratumumab)
* Patients must have Creatinine Clearance above 30 mL/min on the Day 1 of trial
* Patients must have given informed consent to participate in trial.

Exclusion Criteria:

* Contraindication to the use of one of the study drug/vaccines (including known hypersensitivity)
* Creatinine Clearance below 30 mL/min on the Day 1 of trial
* Psychiatric disorder or unable to understand or to follow the protocol directions
* Active bacterial, viral, fungal or protozoal infection on the Day 1 of trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically/radiologically confirmed pneumonia and episodes of febrile neutropenia during one year period after initiation of novel agents. | One year

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | One year
  Data on Common Terminology Criteria for Adverse Events (CTCAE v4.0) will be collected via questionnaires. Measurement data will be aggregated in electronic platform to characterize the frequency, severity and interference of symptomatic treatment toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly Uss, MD/PhD, Study Chair — Minsk Scientific Practical Center of Surgery, Transplantation and Hematology, Belarus
Locations (1):
- Minsk Scientific Practical Center of Surgery, Transplantation and Hematology, Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wallington-Beddoe CT, Pitson SM. Novel therapies for multiple myeloma. Aging (Albany NY). 2017 Aug 28;9(8):1857-1858. doi: 10.18632/aging.101284. No abstract available. PMID 28854147
- [Background] Satlin MJ, Vardhana S, Soave R, Shore TB, Mark TM, Jacobs SE, Walsh TJ, Gergis U. Impact of Prophylactic Levofloxacin on Rates of Bloodstream Infection and Fever in Neutropenic Patients with Multiple Myeloma Undergoing Autologous Hematopoietic Stem Cell Transplantation. Biol Blood Marrow Transplant. 2015 Oct;21(10):1808-14. doi: 10.1016/j.bbmt.2015.06.017. Epub 2015 Jul 3. PMID 26150022
- [Background] Jung SH, Kang SJ, Jang HC, Ahn JS, Yang DH, Lee SS, Kim YK, Kim HJ, Lee JJ. Effect of levofloxacin prophylaxis for prevention of severe infections in multiple myeloma patients receiving bortezomib-containing regimens. Int J Hematol. 2014 Nov;100(5):473-7. doi: 10.1007/s12185-014-1672-1. Epub 2014 Sep 12. PMID 25212681
- [Background] Cordonnier C, Ljungman P, Juergens C, Maertens J, Selleslag D, Sundaraiyer V, Giardina PC, Clarke K, Gruber WC, Scott DA, Schmoele-Thoma B; 3003 Study Group. Immunogenicity, safety, and tolerability of 13-valent pneumococcal conjugate vaccine followed by 23-valent pneumococcal polysaccharide vaccine in recipients of allogeneic hematopoietic stem cell transplant aged >/=2 years: an open-label study. Clin Infect Dis. 2015 Aug 1;61(3):313-23. doi: 10.1093/cid/civ287. Epub 2015 Apr 13. PMID 25870329
- [Result] Stoma I, Karpov I, Iskrov I, Lendina I, Uss A. Clinical efficacy of pneumococcal vaccination in multiple myeloma patients on novel agents: Results of a prospective clinical study. Vaccine. 2020 Jun 19;38(30):4713-4716. doi: 10.1016/j.vaccine.2020.05.024. Epub 2020 May 14. PMID 32418789
- [Derived] Zorger AM, Hirsch C, Baumann M, Feldmann M, Brockelmann PJ, Mellinghoff S, Monsef I, Skoetz N, Kreuzberger N. Vaccines for preventing infections in adults with haematological malignancies. Cochrane Database Syst Rev. 2025 May 21;5(5):CD015530. doi: 10.1002/14651858.CD015530.pub2. PMID 40396505